CLINICAL TRIAL: NCT06491017
Title: Effects of Mechanical Insufflation-Exsufflation With Optimized Settings on Suctioned Wet Mucus Volume During Invasive Ventilation
Brief Title: Effects of Mechanical Insufflation-Exsufflation With Optimized Settings on Wet Mucus Volume During Invasive Ventilation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Joan-Daniel Martí Romeu, Principal Investigator, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HCB/2023/1101
Record Dates: First submitted 2024-02-15; First posted 2024-07-08 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Mucus Retention; Mechanical Ventilation Complication
Keywords: Mechanical insufflation-exsufflation; Physiotherapy; Mucus retention; mechanical ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MI-E intervention protocol (Experimental): The optimized MI-E setting will consist of in-expiratory pressures defined during the previous short-period test to achieve inspiratory volumes of ≥1 liter and PEF ≥80 L/min
  Interventions: Device: MI-E Intervention protocol
- Standard MI-E setting (Active Comparator): The standard MI-E setting will consist of in-expiratory pressures of +40/-40 cmH2O, medium inspiratory flow, with 3 seconds and 2 seconds of in-expiratory time, respectively, and 1-second pause
  Interventions: Device: Standard MI-E setting

INTERVENTIONS:
Device: MI-E Intervention protocol — The endotracheal tube cuff will be inflated to 40 cmH2O and MI-E device will be used to deliver MI-E in automatic mode, with 4 sets of 5 respiratory cycles each and a 1-minute interval between each set.
  Before initiation of the MI-E intervention protocol, the investigators will carry out a short-period test to find the appropriate MI-E settings to achieve inspiratory volumes of ≥1 liter and PEF ≥80 L/min. Concretely, inspiratory and expiratory time will always be set at 4 seconds and 2 seconds, respectively, and inspiratory flow will always be in slow mode. Once the appropriate inspiratory pressure will be found, the expiratory pressure will be initially set to exceed in 30 cmH2O the inspiratory pressure and, if required, this will be increased by 5 cmH2O until achieving a PEF ≥80 L/min with a maximum expiratory pressure of 70 cmH2O.
  Arms: MI-E intervention protocol
Device: Standard MI-E setting — Cough Assist E70 device (Philips Respironics, USA, Andover, Massachusetts) will be used to deliver MI-E in automatic mode, with 4 sets of 5 respiratory cycles each and a 1-minute interval between each set. During the 1-minute pause between sets, the patient will be reconnected to the ventilator to avoid desaturation and de-recruitment during procedures. PEEP will remain stable during the protocol.
  The standard MI-E setting will consist of in-expiratory pressures of +40/-40 cmH2O, medium inspiratory flow, with 3 seconds and 2 seconds of in-expiratory time, respectively, and 1-second pause.
  Arms: Standard MI-E setting

SUMMARY:
Retention of airway secretions is a frequent complication in critically ill patients requiring invasive mechanical ventilation (MV).This complication is often due to excessive secretion production and ineffective secretion clearance.

Mechanical insufflator-exsufflator (MI-E) is a respiratory physiotherapy technique that aims to assist or simulate a normal cough by using an electro-mechanical dedicated device. A positive airway pressure is delivered to the airways, in order to hyperinflate the lungs, followed by a rapid change to negative pressure that promotes a rapid exhalation and enhances peak expiratory flows.

However, there is no consensus on the best MI-E settings to facilitate secretion clearance in these patients. Inspiratory and expiratory pressures of ±40 cmH2O and inspiratory-expiratory time of 3 and 2 seconds, respectively, are often used as a standard for MI-E programming in the daily routine practice, but recent laboratory studies have shown significant benefits when MI-E setting is optimized to promote an expiratory flow bias.

The investigators designed this study to compare the effects of MI-E with an optimized setting versus a standard setting on the wet volume of suctioned sputum in intubated critically ill patients on invasive MV for more than 48 hours.

DETAILED DESCRIPTION:
Retention of airway secretions is a frequent complication in critically ill patients requiring invasive mechanical ventilation (MV). This complication is often due to excessive secretion production and ineffective secretion clearance. One of the main causes is the presence of an endotracheal tube (ETT) which has been shown to decrease mucociliary clearance and hinders the generation of adequate peak expiratory flows when coughing. Other factors such as suboptimal airway humidification, inspiratory flow bias, semi-recumbent position, prolonged immobilization and respiratory muscles weakness further impair sputum clearance. Mucus retention may impede optimal gas exchange, and lead to atelectasis, increased work of breathing, bacterial colonization and development of pulmonary infections, prolonging the need for MV. These conditions, added to initial factors, increase morbidity and mortality in critically ill patients, making secretion clearance an essential factor for patients' prognosis.

Secretion removal techniques, such as, manual or mechanical hyperinflations, chest vibrations or expiratory rib cage compressions, prior to suctioning, are commonly used by physiotherapists in intensive care units (ICU). However, the evidence assessing respiratory physiotherapy techniques in critically ill patients is scant and sometimes inconsistent, making it difficult to extrapolate the results and standardize the clinical practice. Moreover, the execution of these techniques often differs among professionals based on their experience, training, and resources availability.

Mechanical insufflator-exsufflator (MI-E) is a respiratory physiotherapy technique that aims to assist or simulate a normal cough by using an electro-mechanical dedicated device. A positive airway pressure is delivered to the airways, in order to hyperinflate the lungs, followed by a rapid change to negative pressure that promotes a rapid exhalation and enhances peak expiratory flows. MI-E is commonly used in patients with ineffective cough mainly due to respiratory pump failure (i.e: neuromuscular patients), and has been proposed in recent years as a technique with great potential to non-invasively clear secretions in the critically ill. Indeed, recent studies have evaluated safety and efficacy of MI-E in intubated critically ill patients with promising results and no associated adverse events. However, there is no consensus on the best MI-E settings to facilitate secretion clearance in these patients. Inspiratory and expiratory pressures of ±40 cmH2O and inspiratory-expiratory time of 3 and 2 seconds, respectively, are often used as a standard for MI-E programming in the daily routine practice, but recent laboratory studies have shown significant benefits when MI-E setting is optimized to promote an expiratory flow bias. For instance, Volpe et al. achieved significant differences in artificial mucus displacement when inspiratory flows were lowered, inspiratory time was increased to 4 seconds, and expiratory flow bias was enhanced by increasing the expiratory pressure over the inspiratory pressure. More recently, evidence from a swine model confirmed the improvement in mucus movement velocity when expiratory pressure was enhanced to increase the difference between inspiratory and expiratory pressures (i.e: +40/-70cmH2O). Importantly, increased inspiratory pressures should be avoided to prevent movement of mucus toward the lungs and potential associated detrimental effects such as alveolar damage or hemodynamic impairment.

The investigators designed this study to compare the effects of MI-E with an optimized setting versus a standard setting on the wet volume of suctioned sputum in intubated critically ill patients on invasive MV for more than 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18yo).
* Endotracheal intubation and invasive mechanical ventilation for > 48h and active humidification for > 24h.
* Richmond Agitation-Sedation Scale -3 to -5.
* Signed informed consent.

Exclusion Criteria:

* Patients with hemodynamic instability (MAP < 60 or > 110, Heart Rate < 50 or > 130, new onset arrhythmias), respiratory instability (PEEP > 12cmH2O, SpO2 < 90% or fraction of inspired oxygen (FiO2) > 60%).
* Undrained pneumothorax/pneumomediastinum.
* Unstable intracranial pressure (ICP > 20mmHg or MAP < 60).
* Severe bronchospasm.
* Post cardiothoracic surgical patients.
* Active pulmonary tuberculosis.
* Bronchoesophageal or bronchopleural fistulas.
* Prone position.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Wet volume of sputum | Immediately after each intervention
  Airway suctioning will be carried out using an open aspiration procedure, using a 12French catheter connected to a sterile collection container. The suction procedure will be performed according to international guidelines . If necessary, 5 ml of saline solution will be used to rinse the catheter in case of impacted secretions inside the catheter; later this volume will be subtracted from the final volume of secretions, thus obtaining the exact amount of wet sputum.

SECONDARY OUTCOMES:
Respiratory parameters: Inspiratory flow (PIF) | Before and during MI-E interventions, delivered tidal volumes will be recorded, PIF and PEF will be assessed for each insufflation-exsufflation cycle, and the PEF-PIF difference and the PEF:PIF ratio will be calculated
  Flow will be measured with a heated pneumotachograph (Fluxmed GrH monitor MBMED, Buenos Aires, Argentina) inserted between the proximal tip of the endotracheal tube and the Y-piece of the breathing circuit. All signals will be recorded on a personal computer for subsequent analysis with dedicated software (FluxReview software MBMED, Buenos Aires, Argentina)
Respiratory parameters: Peak expiratory flow (PEF) | Before and during MI-E interventions, delivered tidal volumes will be recorded, PIF and PEF will be assessed for each insufflation-exsufflation cycle, and the PEF-PIF difference and the PEF:PIF ratio will be calculated
  Flow will be measured with a heated pneumotachograph (Fluxmed GrH monitor MBMED, Buenos Aires, Argentina) inserted between the proximal tip of the endotracheal tube and the Y-piece of the breathing circuit. All signals will be recorded on a personal computer for subsequent analysis with dedicated software (FluxReview software MBMED, Buenos Aires, Argentina)
Respiratory parameters: difference between PEF-PIF; | Before and during MI-E interventions, delivered tidal volumes will be recorded, PIF and PEF will be assessed for each insufflation-exsufflation cycle, and the PEF-PIF difference and the PEF:PIF ratio will be calculated
  Flow will be measured with a heated pneumotachograph (Fluxmed GrH monitor MBMED, Buenos Aires, Argentina) inserted between the proximal tip of the endotracheal tube and the Y-piece of the breathing circuit. All signals will be recorded on a personal computer for subsequent analysis with dedicated software (FluxReview software MBMED, Buenos Aires, Argentina)
Respiratory parameters: PEF:PIF ratio | Before and during MI-E interventions, delivered tidal volumes will be recorded, PIF and PEF will be assessed for each insufflation-exsufflation cycle, and the PEF-PIF difference and the PEF:PIF ratio will be calculated
  Flow will be measured with a heated pneumotachograph (Fluxmed GrH monitor MBMED, Buenos Aires, Argentina) inserted between the proximal tip of the endotracheal tube and the Y-piece of the breathing circuit. All signals will be recorded on a personal computer for subsequent analysis with dedicated software (FluxReview software MBMED, Buenos Aires, Argentina)
Pulmonary mechanics parameters: Static Compliance (Cst) | Airway pressures will be recorded before, immediately after MI-E intervention, after endotracheal suctioning, and 1h after endotracheal suctioning. Respiratory system compliance and airway resistance will be calculated using standard formulas.
  Pressure signals will be measured with a heated pneumotachograph (Fluxmed GrH monitor MBMED, Buenos Aires, Argentina) inserted between the proximal tip of the endotracheal tube and the Y-piece of the breathing circuit. All signals will be recorded on a personal computer for subsequent analysis with dedicated software (FluxReview software MBMED, Buenos Aires, Argentina)
Pulmonary mechanics parameters: Airway resistance (Raw) | Airway pressures will be recorded before, immediately after MI-E intervention, after endotracheal suctioning, and 1h after endotracheal suctioning. Respiratory system compliance and airway resistance will be calculated using standard formulas.
  Pressure signals will be measured with a heated pneumotachograph (Fluxmed GrH monitor MBMED, Buenos Aires, Argentina) inserted between the proximal tip of the endotracheal tube and the Y-piece of the breathing circuit. All signals will be recorded on a personal computer for subsequent analysis with dedicated software (FluxReview software MBMED, Buenos Aires, Argentina)
Hemodynamics values: Heart rate | Before, immediately after MI-E interventions and after endotracheal suctioning.
  Hemodynamics parameters will be recorder from the patient's monitor.
Hemodynamics values: Mean arterial pressure | Before, immediately after MI-E interventions and after endotracheal suctioning.
  Hemodynamics parameters will be recorded from the patient's monitor.
Gas exchange: Arterial blood gas analysis | Before, immediately after endotracheal suctioning and 1 hour after interventions.
  Parameters will be recorded from the patient's monitor arterial blood gas analysis.
Gas exchange: Pulseoximeter oxygen saturation (SpO2) | Before, immediately after endotracheal suctioning and 1 hour after interventions.
  Parameters will be recorded from patient's pulseoximetry.
Adverse events | During the intervention/procedure and immediately after the intervention/procedure.
  All adverse events that force the interruption of the interventions will be recorded. Reasons to stop MI-E will be haemodynamic instability, severe desaturation, structural damage caused to the airway (i.e. pneumothorax), airway obstruction or difficulty in correct ventilation of the patient.
Numbers of participants with adverse events | During the intervention/procedure and immediately after the intervention/procedure.
  Relationship between the participants who have reported adverse effects and the number of adverse effects in the study.

OTHER OUTCOMES:
Demographic variables: Age | Through study completion
  Age will be collected from the medical record. Age, gender, weight, BMI, height, days of intubation and reason for ICU admission will be collected from the medical record at patient's inclusion.
Demographic variables: Gender | Through study completion, an average of 2 years.
  Gender will be collected from the medical record. Age, gender, weight, BMI, height, days of intubation and reason for ICU admission will be collected from the medical record at patient's inclusion.
Demographic variables: Weight | Through study completion, an average of 2 years.
  Weight (kilograms) will be collected from the medical record. Age, gender, weight, BMI, height, days of intubation and reason for ICU admission will be collected from the medical record at patient's inclusion.
Demographic variables: BMI | Through study completion, an average of 2 years.
  BMI (kg/m^2) will be collected from the medical record. Age, gender, weight, BMI, height, days of intubation and reason for ICU admission will be collected from the medical record at patient's inclusion.
Demographic variables: Height | Through study completion, an average of 2 years.
  Height (meters) will be collected from the medical record. Age, gender, weight, BMI, height, days of intubation and reason for ICU admission will be collected from the medical record at patient's inclusion.
Demographic variables: Days of intubation | Through study completion, an average of 2 years.
  Days of intubation will be collected from the medical record. Age, gender, weight, BMI, height, days of intubation and reason for ICU admission will be collected from the medical record at patient's inclusion.
Demographic variables: Reason for ICU admission | Through study completion, an average of 2 years.
  Reason for ICU admission will be collected from the medical record. Age, gender, weight, BMI, height, days of intubation and reason for ICU admission will be collected from the medical record at patient's inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Daniel Martí, PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Konrad F, Schreiber T, Brecht-Kraus D, Georgieff M. Mucociliary transport in ICU patients. Chest. 1994 Jan;105(1):237-41. doi: 10.1378/chest.105.1.237. PMID 8275739
- [Background] Sackner MA, Hirsch J, Epstein S. Effect of cuffed endotracheal tubes on tracheal mucous velocity. Chest. 1975 Dec;68(6):774-7. doi: 10.1378/chest.68.6.774. PMID 1192854
- [Background] Gal TJ. Effects of endotracheal intubation on normal cough performance. Anesthesiology. 1980 Apr;52(4):324-9. doi: 10.1097/00000542-198004000-00008. PMID 7362053
- [Background] Kilgour E, Rankin N, Ryan S, Pack R. Mucociliary function deteriorates in the clinical range of inspired air temperature and humidity. Intensive Care Med. 2004 Jul;30(7):1491-4. doi: 10.1007/s00134-004-2235-3. Epub 2004 Mar 16. PMID 15024566
- [Background] American Association for Respiratory Care; Restrepo RD, Walsh BK. Humidification during invasive and noninvasive mechanical ventilation: 2012. Respir Care. 2012 May;57(5):782-8. doi: 10.4187/respcare.01766. PMID 22546299
- [Background] Li Bassi G, Zanella A, Cressoni M, Stylianou M, Kolobow T. Following tracheal intubation, mucus flow is reversed in the semirecumbent position: possible role in the pathogenesis of ventilator-associated pneumonia. Crit Care Med. 2008 Feb;36(2):518-25. doi: 10.1097/01.CCM.0000299741.32078.E9. PMID 18176317
- [Background] Wu MF, Wang TY, Chen DS, Hsiao HF, Hu HC, Chung FT, Lin TY, Lin SM. The effects of mechanical insufflation-exsufflation on lung function and complications in cardiac surgery patients: a pilot study. J Cardiothorac Surg. 2021 Dec 9;16(1):350. doi: 10.1186/s13019-021-01738-x. PMID 34886881
- [Background] Kuroiwa R, Tateishi Y, Oshima T, Inagaki T, Furukawa S, Takemura R, Kawasaki Y, Murata A. Mechanical Insufflation-exsufflation for the Prevention of Ventilator-associated Pneumonia in Intensive Care Units: A Retrospective Cohort Study. Indian J Crit Care Med. 2021 Jan;25(1):62-66. doi: 10.5005/jp-journals-10071-23508. PMID 33603304
- [Background] Pneumatikos IA, Dragoumanis CK, Bouros DE. Ventilator-associated pneumonia or endotracheal tube-associated pneumonia? An approach to the pathogenesis and preventive strategies emphasizing the importance of endotracheal tube. Anesthesiology. 2009 Mar;110(3):673-80. doi: 10.1097/ALN.0b013e31819868e0. PMID 19212256
- [Background] Shapiro M, Wilson RK, Casar G, Bloom K, Teague RB. Work of breathing through different sized endotracheal tubes. Crit Care Med. 1986 Dec;14(12):1028-31. doi: 10.1097/00003246-198612000-00007. PMID 3780244
- [Background] Branson RD. Secretion management in the mechanically ventilated patient. Respir Care. 2007 Oct;52(10):1328-42; discussion 1342-7. PMID 17894902
- [Background] Martinez-Alejos R, Marti JD, Li Bassi G, Gonzalez-Anton D, Pilar-Diaz X, Reginault T, Wibart P, Ntoumenopoulos G, Tronstad O, Gabarrus A, Quinart A, Torres A. Effects of Mechanical Insufflation-Exsufflation on Sputum Volume in Mechanically Ventilated Critically Ill Subjects. Respir Care. 2021 Sep;66(9):1371-1379. doi: 10.4187/respcare.08641. Epub 2021 Jun 8. PMID 34103385
- [Background] Rose L, McKim D, Leasa D, Nonoyama M, Tandon A, Kaminska M, O'Connell C, Loewen A, Connolly B, Murphy P, Hart N, Road J. Monitoring Cough Effectiveness and Use of Airway Clearance Strategies: A Canadian and UK Survey. Respir Care. 2018 Dec;63(12):1506-1513. doi: 10.4187/respcare.06321. Epub 2018 Sep 11. PMID 30206128
- [Background] Goni-Viguria R, Yoldi-Arzoz E, Casajus-Sola L, Aquerreta-Larraya T, Fernandez-Sangil P, Guzman-Unamuno E, Moyano-Berardo BM. Respiratory physiotherapy in intensive care unit: Bibliographic review. Enferm Intensiva (Engl Ed). 2018 Oct-Dec;29(4):168-181. doi: 10.1016/j.enfi.2018.03.003. Epub 2018 Jun 15. English, Spanish. PMID 29910086
- [Background] Swingwood E, Tume L, Cramp F. A survey examining the use of mechanical insufflation-exsufflation on adult intensive care units across the UK. J Intensive Care Soc. 2020 Nov;21(4):283-289. doi: 10.1177/1751143719870121. Epub 2019 Sep 5. PMID 34093728
- [Background] Sanchez-Garcia M, Santos P, Rodriguez-Trigo G, Martinez-Sagasti F, Farina-Gonzalez T, Del Pino-Ramirez A, Cardenal-Sanchez C, Busto-Gonzalez B, Requesens-Solera M, Nieto-Cabrera M, Romero-Romero F, Nunez-Reiz A. Preliminary experience on the safety and tolerability of mechanical "insufflation-exsufflation" in subjects with artificial airway. Intensive Care Med Exp. 2018 Apr 3;6(1):8. doi: 10.1186/s40635-018-0173-6. PMID 29616357
- [Background] Volpe MS, Naves JM, Ribeiro GG, Ruas G, Amato MBP. Airway Clearance With an Optimized Mechanical Insufflation-Exsufflation Maneuver. Respir Care. 2018 Oct;63(10):1214-1222. doi: 10.4187/respcare.05965. Epub 2018 Jul 17. PMID 30018177
- [Background] Volpe MS, Guimaraes FS, Morais CC. Airway Clearance Techniques for Mechanically Ventilated Patients: Insights for Optimization. Respir Care. 2020 Aug;65(8):1174-1188. doi: 10.4187/respcare.07904. PMID 32712584
- [Background] Rose L, Adhikari NK, Leasa D, Fergusson DA, McKim D. Cough augmentation techniques for extubation or weaning critically ill patients from mechanical ventilation. Cochrane Database Syst Rev. 2017 Jan 11;1(1):CD011833. doi: 10.1002/14651858.CD011833.pub2. PMID 28075489
- [Background] Benditt JO. Mechanical Insufflation-Exsufflation: More Than Just Cough Assist. Respir Care. 2018 Aug;63(8):1076-1077. doi: 10.4187/respcare.06439. No abstract available. PMID 30045899
- [Background] Chatwin M, Simonds AK. Long-Term Mechanical Insufflation-Exsufflation Cough Assistance in Neuromuscular Disease: Patterns of Use and Lessons for Application. Respir Care. 2020 Feb;65(2):135-143. doi: 10.4187/respcare.06882. Epub 2019 Nov 5. PMID 31690614
- [Background] Ferreira de Camillis ML, Savi A, Goulart Rosa R, Figueiredo M, Wickert R, Borges LGA, Galant L, Teixeira C. Effects of Mechanical Insufflation-Exsufflation on Airway Mucus Clearance Among Mechanically Ventilated ICU Subjects. Respir Care. 2018 Dec;63(12):1471-1477. doi: 10.4187/respcare.06253. Epub 2018 Jul 17. PMID 30018175
- [Background] Marti JD, Martinez-Alejos R, Pilar-Diaz X, Yang H, Pagliara F, Battaglini D, Meli A, Yang M, Bobi J, Rigol M, Tronstad O, Volpe MS, Passos Amato MB, Bassi GL, Torres A. Effects of Mechanical Insufflation-Exsufflation With Different Pressure Settings on Respiratory Mucus Displacement During Invasive Ventilation. Respir Care. 2022 Dec;67(12):1508-1516. doi: 10.4187/respcare.10173. Epub 2022 Aug 30. PMID 36041752